CLINICAL TRIAL: NCT05715151
Title: Impact of Externally Facilitated Continuous Quality Improvement Cohorts on Advanced Access to Support Primary Healthcare Teams
Brief Title: Continuous Quality Improvement Cohorts on Advanced Access
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: Isabelle Gaboury (Unknown); Mike Green (Unknown); Tara Kiran (Unknown); Janusz Kaczorowski (Unknown); Maude Laberge (Unknown)
Responsible Party: Principal Investigator, Mylaine Breton, Associate Professor, Department of Community Health Sciences, Université de Sherbrooke
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MP-04-2022-696
Record Dates: First submitted 2022-12-21; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Primary Health Care
Keywords: Advanced Access; Primary Health Care; Quality improvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CQI intervention (Experimental): The proposed CQI cohort consists of three activities carried out iteratively until the improvement objectives are achieved.
  Interventions: Other: CQI intervention
- Audit and feedback (Active Comparator): Clinics in the control group will receive feedback on six key AA indicators, patients reported experience about access and selected AA processes.
  Interventions: Other: Audit and Feedback

INTERVENTIONS:
Other: CQI intervention — Activity 1: Reflective sessions and problem prioritisation. Activity 2: PDSA cycles. Activity 3: Group mentoring.
  Arms: CQI intervention
Other: Audit and Feedback — Audit and Feedback on six key AA indicators, patients reported experience about access and selected AA processes.
  Arms: Audit and feedback

SUMMARY:
The goal of this clinical trial is to compare the implementation and effects of CQI cohorts on AA for PHC clinics. The main questions it aims to answer are to assess the effectiveness of CQI cohorts on AA outcomes.

DETAILED DESCRIPTION:
SIGNIFICANCE AND PURPOSE: Timely access to primary healthcare is one cornerstone of strong primary healthcare. Across Canada, timely access remains a significant challenge. One of the most highly recommended models around the world to improve timely access is advanced access (AA). Over the last two decades, AA has become increasingly popular in Canada. AA model has been widely promoted by the College of Family Physicians of Canada and several other provincial organizations and professional associations. Some tools to support the implementation of AA to PHC providers and practices have been developed such as workbook by Health Quality Ontario and Doctor of BC. However, those tools are important assets to initiate a reflection to improve, they are often not sufficient. Eight PHC teams interested in improving and expanding the implementation of AA have been coached through several PDSA cycles. However, the personalized support model used is very demanding in terms of capacity and resources. These findings guided the research team in developing and evaluating a Continuous Quality Improvement (CQI) Cohort program on advanced access to support Primary healthcare (PHC) teams.This study aims to develop knowledge on an externally facilitated CQI pan-Canadian cohort program that could potentially be transferred to provincial organizations or professional associations wishing to support clinics in quality improvement projects.

OBJECTIVE: Assess the effectiveness of CQI cohorts on AA outcomes.

QI INTERVENTION PROGRAM: PHC teams will participate in an externally facilitated CQI program focusing on AA. The proposed program consists of cycle of three key activities; 1) Interprofessional reflective sessions and need prioritization, 2) Group mentoring and PDSA Cycles and 3) Cohort cross-learning exchange opportunities.

METHODS: This study will be based on the cluster-controlled trial of a CQI program of PHC teams on AA. 48 PHC teams from Quebec will participate to the externally facilitated CQI cohort intervention. Volunteer clinics from the intervention regions will receive the CQI intervention for 18 months. Intervention clinics will be matched to PHC clinics located in other regions to compose the control group. The match will be based on the clinic level (1 to 10, based on the number of patients registered and services offered. Clinics in the control group will receive an audit on a selection of AA indicators and will be offered the intervention 12 to 18 months following their recruitment. Data collection and analysis will include quantitative data based on a comprehensive assessment of both AA processes and outcomes. These will be measured through a self-reflective survey for PHC team members, EMR data and patients related outcomes questionnaire on access. Qualitative data based on semi-structured interviews with key stakeholders, observations of the CQI activities and analysis of plans of action of documents plan of action will take place.

ELIGIBILITY:
Inclusion criteria:

* Clinics must offer interprofessional care.
* At least 50 % of all team members should accept to take part in the study.

Exclusion criteria:

* Solo Practice Physicians
* Physician-nurse only model

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
3rd next available appointment (weekly) | 18 month
  Delay before the 3rd next available appointment. The 3rd next available appointment is used (rather than the 1st or 2nd) to decrease variation.
Percent of relational continuity (monthly) | 18 month
  Total number of medical consultations with a patient's attached family physician (or specialised nurse) out of the total number of consultations with any family physician (or specialised nurse) from the clinic. Evaluates relational continuity between the provider and their registered patients.

SECONDARY OUTCOMES:
Percent of 48-hour open slots (weekly) | 18 month
  Proportion of appointments available in the next 48 hours. Provides an overview of the provider's ability to respond to urgent care demands.
Use of walk-in (monthly) | 18 month
  Proportion of walk-in visits by registered patients to each professional.
Proportion of multidisciplinary involvement (monthly) | 18 month
  Evaluates the proportion of involvement of different types of providers (social workers, nurses, pharmacists, etc.) with registered patients.
Discontinuity for chronic patients (monthly) | 18 month
  Proportion of chronic patients without any consultations within the last 12 months.
3rd next available appointment (weekly) | 12 month
  Delay before the 3rd next available appointment. The 3rd next available appointment is used (rather than the 1st or 2nd) to decrease variation.
Percent of relational continuity (monthly) | 12 month
  Total number of medical consultations with a patient's attached family physician (or specialised nurse) out of the total number of consultations with any family physician (or specialised nurse) from the clinic. Evaluates relational continuity between the provider and their registered patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mylaine Breton, PhD, Principal Investigator — Université de Sherbrooke
Locations (18):
- Canada (18):
  - CISSS de la Gaspésie, Gaspé, Quebec
  - CISSS de l'Outaouais, Gatineau, Quebec
  - CISSS de Lanaudière, Joliette, Quebec
  - CISSS de Laval, Laval, Quebec
  - CISSS de Chaudière-Appalaches, Lévis, Quebec
  - CIUSSS de Montérégie-Centre, Longueuil, Quebec
  - CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal, Quebec
  - CIUSSS de l'Ouest-de-l'Île-de-Montréal, Montreal, Quebec
  - CIUSSS du Centre-Ouest-de-l'Île-de-Montréal, Montreal, Quebec
  - CIUSSS du Centre-Sud-de-l'Île-de-Montréal, Montreal, Quebec
  - CIUSSS du Nord-de-l'Île-de-Montréal, Montreal, Quebec
  - CISSS de l'Abitibi-Témiscamingue, Rouyn-Noranda, Quebec
  - CISSS de la Montérégie-Ouest, Saint-Hubert, Quebec
  - CISSS de la Montérégie-Est, Saint-Hyacinthe, Quebec
  - CISSS des Laurentides, Saint-Jérôme, Quebec
  - CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec
  - CIUSSS de la Mauricie et Centre-du-Québec, Trois-Rivières, Quebec
  - CIUSSS de la Capitale-Nationale, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breton M, Gaboury I, Martin E, Green ME, Kiran T, Laberge M, Kaczorowski J, Ivers N, Deville-Stoetzel N, Bordeleau F, Beaulieu C, Descoteaux S. Impact of externally facilitated continuous quality improvement cohorts on Advanced Access to support primary healthcare teams: protocol for a quasi-randomized cluster trial. BMC Prim Care. 2023 Apr 11;24(1):97. doi: 10.1186/s12875-023-02048-y. PMID 37038126